CLINICAL TRIAL: NCT00949091
Title: A Phase 1, Double-Blind, Randomized, Placebo-Controlled, Sequential, Multiple Ascending-Dose Study to Evaluate the Pharmacokinetics and Pharmacodynamics of TAK-875 in Subjects With Type 2 Diabetes
Brief Title: Pharmacokinetics and Pharmacodynamics of TAK-875 in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sr. VP, Clinical Science, Takeda Global Research & Development Center, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: TAK-875_102; U1111-1114-2888 (Registry Identifier: WHO)
Record Dates: First submitted 2009-07-28; First posted 2009-07-30 (Estimated); Last update posted 2010-06-11 (Estimated); Status verified 2010-06

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus, Non Insulin Dependent; Diabetes Mellitus, Type II; Type 2 Diabetes Mellitus; Drug Therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — TAK-875

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: TAK-875

INTERVENTIONS:
Drug: TAK-875 — Randomized, multiple ascending-dose sequence over 14 consecutive days to include the following:
  TAK-875 25 mg tablets, orally
  TAK-875 50 mg tablets, orally
  TAK-875 100 mg tablets, orally
  TAK-875 200 mg tablets, orally
  TAK-875 400 mg tablets, orally
  TAK-875 placebo-matching tablets, orally.

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of multiple ascending-doses of TAK-875 in subjects with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
TAK-875 is being developed as an adjunct to diet and exercise to improve glycemic control in patients with type 2 diabetes mellitus. Nonclinical data suggest that TAK-875 stimulates insulin secretion only at elevated blood glucose levels, with the potential for low hypoglycemic side effects.

The purpose of this phase 1, multiple ascending-dose study is to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of once daily oral doses of TAK-875 for 14 days in subjects with type 2 diabetes mellitus.

Participants will be housed for a total of 8 consecutive overnight stays in the clinic, and will undergo oral glucose tolerance tests and standardized meal tests with multiple blood sampling throughout their clinic stay.

ELIGIBILITY:
Inclusion Criteria:

* Participants with type 2 diabetes who are newly diagnosed, managed with diet and exercise alone, or taking up to 2 oral antidiabetic agents (except thiazolidinediones) and willing to discontinue the antidiabetic medication(s) 2 weeks prior to randomization.
* Meets one of the following glycosylated hemoglobin criteria (diagnosis must be based on current American Diabetes Association criteria) at Screening:

  * If treatment naïve, should have a glycosylated hemoglobin concentration greater than or equal to 6.5% and less than or equal to 10.0%.
  * If on a single antidiabetic agent (stable dose for at least 28 days), should have a glycosylated hemoglobin greater than or equal to 6% and less than or equal to 9.5%.
  * If on a combination of up to 2 antidiabetic agents (stable doses for at least 28 days), should have a glycosylated hemoglobin greater than or equal to 6% and less than or equal to 9.0%.
* Has fasting plasma glucose greater than 126 mg/dL and less than 260 mg/dL if not on any antidiabetic medication, or less than 220 mg/dL if on any single antidiabetic agent, and less than 200 mg/dL if on any combination of 2 oral antidiabetic agents at Screening.
* Has fasting C-peptide concentration greater than or equal to 0.8 ng/mL at Screening.
* Weighs at least 50 kg (110 lb) and has a body mass index between 18 and 40 kg/m2, inclusive at Screening.
* Has not received treatment with weight-loss drugs within the 3 months prior to Screening.
* Has a systolic blood pressure less than or equal to 160 mm Hg and a diastolic blood pressure of less than or equal to 100 mm Hg at Screening and at Check-in (Day -2).
* Female participant is not of child-bearing potential (ie, surgically sterile [hysterectomy, bilateral oophorectomy, or 2 years post-tubal ligation] or postmenopausal [2 years since last menses]).
* Is able and willing to monitor blood glucose concentrations with a home glucose monitor during the Washout Interval and record results in the daily diary.
* Has negative test results at Screening and Check-in for selected substances of abuse, including alcohol and cotinine.
* Has Screening and Check-in clinical laboratory evaluations [including fasting clinical chemistry, hematology, and complete urinalysis (excluding glucose results)] within the reference range for the testing laboratory, unless the investigator deems the out-of-range results to be not clinically significant.
* Has negative test results for hepatitis B surface antigen and antibody to hepatitis C virus, and no known history of human immunodeficiency virus.
* Is willing to refrain from strenuous exercise from 72 hours before Check-in and throughout the study.
* Is considered by the investigator to be in a good health (other than being diabetic) as determined during the medical history review, physical examination findings, electrocardiogram and vital sign results, and clinical laboratory evaluations.
* Has creatinine clearance greater than 60 mL/min at Screening and Check-in.

Exclusion Criteria:

* Has a history of abdominal surgery (except laparoscopic cholecystectomy or uncomplicated appendectomy), thoracic, or nonperipheral vascular surgery within 6 months prior to Check-in.
* Has a known hypersensitivity to TAK-875, or other related compounds.
* Has a history of cardiac arrhythmia, systolic dysfunction congestive heart failure, angina, myocardial ischemia or infarction, or stroke within 1 year prior to Screening, or the presence of an abnormal electrocardiogram that, in the investigator's opinion, is clinically significant.
* Has a history of drug abuse or a history of alcohol abuse within 2 years prior to Screening.
* Has used any tobacco (ie, nicotine) products within 90 days prior to Check-in, and is unwilling to abstain from these products for the duration of the study.
* Has a history of cancer that has not been in remission for at least 5 years prior to the first dose of study drug. This criterion does not apply to basal cell or stage I squamous cell carcinoma of the skin.
* Has an alanine aminotransferase, alkaline phosphatase or aspartate aminotransferase level greater than or equal to 2 times the upper limit normal for the testing laboratory, active liver disease, or jaundice at Screening or Check-in.
* Has a total bilirubin greater than 2 mg/dL at Screening or Check-in.
* Has donated blood or experienced acute blood loss (including plasmapheresis) of greater than 500 mL within 90 days prior to the first dose of study drug.
* Participant is on any insulin treatment.
* The subject has a history of proteinuria greater than 300 mg/day on a 12- or 24-hour urine collection or an albumin/creatinine ratio greater than 300 μg/mg at Screening. If elevated, the subject may be rescreened within 1 week, and may be included in study with agreement between Principal Investigator and the Takeda Global Research and Development Medical Monitor.
* Has a history of any clinically significant retinopathy, which is defined as more than moderate nonproliferative diabetic retinopathy or any stage of proliferative diabetic retinopathy or any history of laser-treated retinopathy.
* Has history of treated or clinically significant peripheral or autonomic neuropathy.
* The subject has a history of ulcerative colitis or Crohn's disease, or has undergone gastric resection.
* The subject has a history of a psychiatric disorder that will affect the subject's ability to participate in the study.
* Has a history of angioedema.
* Had an acute, clinically significant illness within 30 days prior to Check-in, or any other condition or prior therapy that, in the opinion of the investigator, would make the subject unsuitable for the study.
* Participant took or requires the use of any restricted medication or products within the timeframes listed.
* Is participating in another investigational study or has taken any investigational drug within 30 days prior to Check-in.
* Has poor venous access.
* Has been randomized in a previous TAK-875 study within 6 months prior to the first dose of study drug.

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-01; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
TAK-875 maximum observed plasma concentration (Cmax) | Day 14
TAK-875 time at which Cmax occurred (Tmax) | Day 14
TAK-875 area under the plasma concentration-time curve from time 0 to time tau, where tau is the length of a dosing interval AUC(0-tau) | Day 14
TAK-875 renal clearance (CLr) | Day 14
TAK-875 metabolite (M-I) Cmax | Day 14
TAK-875 M-I Tmax | Day 14
TAK-875 M-I AUC(0-tau) | Day 14
TAK-875 M-I renal clearance CLr | Day 14

SECONDARY OUTCOMES:
TAK-875 Cmax | Day 1
TAK-875 Tmax | Day 1
TAK-875 AUC(0-tau) | Day 1
TAK-875 renal clearance CLr | Day 1
M-I Tmax | Day 1
M-I Cmax | Day 1
M-I AUC(0-tau) | Day 1
M-I renal clearance CLr | Day 1
TAK-875 and M-I Cmax ratio | Day 1
TAK-875 and M-I Cmax ratio | Day 14
TAK-875 and M-I AUC(0-tau) ratio | Day 1
TAK-875 and M-I AUC(0-tau) ratio | Day 14
Percent changes from baseline to Day 14 in mean 4-hour concentration values for plasma glucose | Day 14
Percent changes from baseline to Day 14 in mean 4- hour concentration values for insulin | Day 14
Percent changes from baseline to Day 14 in mean 4- hour concentration values for proinsulin | Day 14
Percent changes from baseline to Day 14 in mean 4- hour concentration values for C-peptide | Day 14
Percent changes from baseline to Day 14 in mean 4- hour concentration values for glucagon | Day 14
Percent changes from baseline to Day 14 in mean 4- hour concentration values for total gastric inhibitory polypeptide (GIP) | Day 14
Percent changes from baseline to Day 14 in mean 4- hour concentration values for total glucagon-like peptide-1 (GLP-1) | Day 14
Percent changes from baseline to Day 14 in mean 24-hour concentration values for plasma glucose | Day 14
Percent changes from baseline to Day 14 in mean 24- hour concentration values for insulin | Day 14
Percent changes from baseline to Day 14 in mean 24- hour concentration values for proinsulin | Day 14
Percent changes from baseline to Day 14 in mean 24- hour concentration values for C-peptide | Day 14
Percent changes from baseline to Day 14 in mean 24- hour concentration values for glucagon | Day 14
Percent changes from baseline to Day 14 in mean 24- hour concentration values for total gastric inhibitory polypeptide (GIP) | Day 14
Percent changes from baseline to Day 14 in mean 24- hour concentration values for total glucagon-like peptide-1 (GLP-1) | Day 14
Absolute changes from baseline to Day 14 in mean 4-hour concentration values for plasma glucose | Day 14
Absolute changes from baseline to Day 14 in mean 4- hour concentration values for insulin | Day 14
Absolute changes from baseline to Day 14 in mean 4- hour concentration values for proinsulin | Day 14
Absolute changes from baseline to Day 14 in mean 4- hour concentration values for C-peptide | Day 14
Absolute changes from baseline to Day 14 in mean 4- hour concentration values for glucagon | Day 14
Absolute changes from baseline to Day 14 in mean 4- hour concentration values for total gastric inhibitory polypeptide (GIP) | Day 14
Absolute changes from baseline to Day 14 in mean 4- hour concentration values for total glucagon-like peptide-1 (GLP-1) | Day 14
Absolute changes from baseline to Day 14 in mean 24-hour concentration values for plasma glucose | Day 14
Absolute changes from baseline to Day 14 in mean 24- hour concentration values for insulin | Day 14
Absolute changes from baseline to Day 14 in mean 24- hour concentration values for proinsulin | Day 14
Absolute changes from baseline to Day 14 in mean 24- hour concentration values for C-peptide | Day 14
Absolute changes from baseline to Day 14 in mean 24- hour concentration values for glucagon | Day 14
Absolute changes from baseline to Day 14 in mean 24- hour concentration values for total gastric inhibitory polypeptide (GIP) | Day 14
Absolute changes from baseline to Day 14 in mean 24- hour concentration values for total glucagon-like peptide-1 (GLP-1) | Day 14
Percent change from baseline to 24-hours post Day 13 dose in homeostasis model assessment of ß-cell function | Day 13
Percent change from baseline to 24-hours post Day 14 dose in homeostasis model assessment of ß-cell function | Day 14
Absolute change from baseline to 24-hours post Day 13 dose in homeostasis model assessment of ß-cell function | Day 13
Absolute change from baseline to 24-hours post Day 14 dose in homeostasis model assessment of ß-cell function | Day 14
Percent change from baseline to Day 14 in insulinogenic index | Day 14
Absolute change from baseline to Day 14 in insulinogenic index | Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda